CLINICAL TRIAL: NCT01086488
Title: A Phase II, Randomized Controlled Trial of Foscan®-Mediated Photodynamic Therapy Versus Brachytherapy in Patients With Recurrent or Persistent Nasopharyngeal Carcinoma
Brief Title: Foscan®-Mediated Photodynamic Therapy Versus Brachytherapy in Patients With Nasopharyngeal Carcinoma
Acronym: FOSCAN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ministry of Health, Malaysia (Other Government)
Responsible Party: Yoke-Yeow Yap, MD, Name/Official Title: Dr. Yap Yoke Yeow
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT 08-03; major research grant (Other: National Medical Research Registry)
Record Dates: First submitted 2010-03-11; First posted 2010-03-15 (Estimated); Last update posted 2011-07-08 (Estimated); Status verified 2011-07

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: recurrent or persistent Nasopharyngeal Carcinoma; treatment of patients with squamous cell carcinoma of the head and neck; Foscan-PDT; Brachytherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Recurrence | interventions — temoporfin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nasopharyngeal Carcinoma (Experimental): A: Experimental B: Active Comparator
  Interventions: Drug: FOSCAN

INTERVENTIONS:
Drug: FOSCAN — Patients will be randomised to one of two treatment groups. The first group of 26 patients will receive 0.1 mg/kg Foscan® at a drug-light interval of 48 hours (2 days). A single surface illumination light dose of 20 J/cm2 fluence rate of 50 mW at 652 nm will be used. The second reference group of 26 patients will be treated by intracavitary brachytherapy

SUMMARY:
Objectives:

Primary objective

- To determine the efficacy of Foscan-PDT compared with Brachytherapy for recurrent or persistent NPC, as determined by macroscopic clinical examination, CT scan and biopsy. The primary endpoint is complete tumour response at 6 months.

Secondary objective:

* To determine the response rates, e.g. presence of tumour on endoscopy, time to progression and overall survival in patients treated with Foscan-PDT compared with brachytherapy
* To determine the quality of life, as derived from the University of Washington Quality of Life questionnaire in patients treated with Foscan-PDT compared with brachytherapy
* To evaluate the safety of Foscan-PDT compared with brachytherapy in terms of adverse events and serious adverse events.

DETAILED DESCRIPTION:
This is a multi-centre, randomized, controlled Phase II study assessing the use of Foscan®-mediated photodynamic therapy versus Brachytherapy in patients with recurrent or persistent nasopharyngeal carcinoma.

The starting point for the PDT arm of the study will be the parameters recommended for the treatment of patients with squamous cell carcinoma of the head and neck. These parameters (drug dose, 0.1 mg/kg Foscan®; drug-light interval, 48 hours; light dose, 20 J/cm2 at 50 mW) have been shown to be effective in a limited number of treatments performed in patients with nasopharyngeal carcinoma.

Patients will be evaluated on a regular basis for 12 weeks following treatment. Patients with a persistent tumour (confirmed histologically, where clinically possible) at 12 weeks following treatment, and in whom adequate clinical assessment of tumour response is possible, may be retreated with Foscan®. A maximum of two Foscan®-PDT treatments may administered to a single patient. Patients will be followed up for up to 24 months following the final Foscan®-PDT treatment.

Study population Any patient with recurrent or persistent nasopharyngeal carcinoma, at least 3 months following a full course of irradiation, is eligible for assessment for enrolment in the study provided that the tumour is less or equal to 15 mm in depth and is accessible for unrestricted illumination using a nasopharyngeal applicator. Diagnosis of cancer will, in the first instance, be made by clinical inspection of the site. The diagnosis must then be confirmed histologically. All patients will have a full assessment and diagnostic workup in accordance with usual departmental practices, including a CT scan of the skull base and neck.

The study centres will keep a log of all patients screened or evaluated for inclusion into the study and will document the reasons why patients were not included or selected.

ELIGIBILITY:
Inclusion Criteria:

Patients will be deemed eligible for inclusion if all the following criteria are met.

* Histologically confirmed local or locoregional recurrent or persistent NPC, [T1-2a, N1-2; M0] at least 3 months following a full course of irradiation
* Discrete tumour, less or equal to 15 mm in depth, which is endoscopically visible and accessible for unrestricted surface illumination using a nasopharyngeal applicator, with no bony invasion
* Patient is 18 - 69 years of age, and legally competent
* Patient has a ECOG performance status ≤2
* Patient is a man or a non-pregnant, non-lactating woman
* Patient, or his legally appointed representative, is able and willing to provide informed consent to participate in the study

Exclusion Criteria:

Patients will not be deemed eligible for inclusion if any of the following criteria apply.

* Elective surgery is planned for within 30 days of administration of Foscan®
* Patient has any disease, which is caused or exacerbated by light, including systemic lupus erythematosus, psoriasis, porphyria, actinic reticuloid or xeroderma pigmentosum
* Patient has been treated within the prior 30 days with a light-activated therapy or other medication that may render the patient photosensitive (e.g., psoralen ultraviolet A-range [PUVA], Accutane)
* Patient has received prior photodynamic therapy to the proposed treatment site within the prior 3 months
* Patient has co-existing ophthalmic disease, which is likely to require slit lamp examination within 30 days following Foscan® administration
* Patient has a known hypersensitivity to temoporfin, or any of the excipients, or to porphyrins
* Patient has a tumour known to be eroding into a major blood vessel in, or adjacent to, the proposed illumination site
* Patient is of childbearing potential and will not use adequate contraceptive protection. Patient should practice strict birth control (oestrogen-containing oral contraceptives or an intrauterine device) throughout the study. Only post-menopausal women (at least 2 years since the onset of the menopause) and women who have had a hysterectomy are exempt from the requirement to use birth control.
* Patient has received treatment with an experimental drug within the prior 30 days
* Patient has received radiotherapy to the head and neck region within the prior 3 months
* Patient is not willing or able to complete the visit requirements of this protocol or adhere to the instructions regarding light exposure

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-09 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint: To determine the efficacy of Foscan-PDT compared with Brachytherapy for recurrent or persistent NPC, as determined by macroscopic clinical examination, CT scan and biopsy. | 12 months

SECONDARY OUTCOMES:
To determine the response rates | 12 months
  To determine the response rates, e.g. presence of tumour on endoscopy, time to progression and overall survival in patients treated with Foscan-PDT compared with brachytherapy. To determine the quality of life. To evaluate the safety of Foscan-PDT compared with brachytherapy in terms of adverse events and serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Yoke Yeow Yap, MD, Principal Investigator — University Putra Malaysia
Locations (5):
- Malaysia (5):
  - Hospital Universiti Sains Malaysia, Kubang Kerian, Kelantan
  - Queen Elizabeth Hospital, Kota Kinabalu, Sabah
  - Universiti Malaysia Sarawak, Kuching, Sarawak
  - Hospital Pulau Pinang, George Town
  - Kuala Lumpur Hospital, Kuala Lumpur

REFERENCES:
- See also: Related Info — http://www.crc.gov.my